CLINICAL TRIAL: NCT01603368
Title: Prophylactic Probiotics to Extremely Low Birth Weight Prematures
Acronym: PROPEL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ostergotland County Council, Sweden (Other)
Collaborators: BioGaia AB (Industry); Ekhaga Foundation, Sweden (Unknown); Medical Research Council of Southeast Sweden (Other Government); University Hospital, Linkoeping (Other); The Swedish Research Council (Other Government); The Swedish Society of Medicine (Other)
Responsible Party: Principal Investigator, Thomas Abrahamsson, MD, PhD, MD, PhD, Neonatologist, Ostergotland County Council, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Dnr 2012/28-31
Record Dates: First submitted 2012-05-18; First posted 2012-05-22 (Estimated); Results first posted 2020-04-27 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Feeding; Difficult, Newborn; Growth Failure; Necrotizing Enterocolitis; Sepsis
Keywords: Probiotics; Lactobacillus reuteri; Prematures; Enteral feeding; Motility; Necrotizing enterocolitis; Sepsis; Weight
MeSH Terms: conditions — Failure to Thrive; Enterocolitis, Necrotizing; Sepsis; Body Weight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactobacillus reuteri (Active Comparator): Lactobacillus reuteri DSM 17938, 125 million bacteria/day
  Interventions: Dietary Supplement: Lactobacillus reuteri
- Placebo (Placebo Comparator): The same oil drops as the active study product but without Lactobacillus reuteri
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri — Oil drops with Lactobacillus reuteri DSM 17938, 125 million bacteria=0.2 ml per day
  Arms: Lactobacillus reuteri
Dietary Supplement: Placebo — Oil drops without Lactobacillus reuteri
  Arms: Placebo

SUMMARY:
Mortality and incidence of severe complications is still high among extremely premature infants. Common causes of severe complications in this population are poor nutrition, necrotizing enterocolitis, and severe infections. Feeding intolerance is also a common problem resulting in prolonged need for intravenous lines and poor nutrition.

The aim of the study is to evaluate whether supplementation with the probiotic bacterium Lactobacillus reuteri DSM 17938 daily to premature infants with extremely low birth weight increases feeding tolerance to breast milk and thereby improves nutrition, increases growth and reduces serious complications and mortality in this population. Beyond this, possible mechanisms underlying these effects will be analyzed in stool, breast milk and blood samples.

DETAILED DESCRIPTION:
RATIONALE Mortality and incidence of severe complications is still high among extremely premature infants. Common causes of severe complications in this population are poor nutrition, necrotizing enterocolitis (NEC), and severe infections. Feeding intolerance is also a common problem resulting in prolonged need for intravenous lines and poor nutrition. There is scientific evidence that dietary supplements with probiotics may have an effect on these manifestations.

Lactobacillus reuteri is a well studied probiotic bacterium that has been tested in several clinical studies in premature infants and older children, and the results of these studies and animal studies suggest that this bacterium may also have an effect on growth and mortality in extremely premature infants. Lactobacillus reuteri reduces colonization with pathogenic microbes, stimulates gastric and intestinal motility and shortens hospital stay in moderately premature infants. In animal models, L. reuteri also induces anti-inflammatory immune responses, reduces the symptoms of inflammatory bowel disease and the incidence of NEC. Administration of L. reuteri also improves the intestinal barrier both in human studies in children and in animal studies. Dietary supplements of L. reuteri to extremely premature infants may therefore improve feeding tolerance and nutrition and reduce the incidence of severe complications in this population.

HYPOTHESIS Premature infants with extremely low birth weight receiving daily supplements of Lactobacillus reuteri DSM 17938 will reach full enteral feeding faster compared with children receiving placebo.

STUDY DESIGN This study will be conducted as a prospective multi-center double blind placebo-controlled study in neonatal intensive care units in Sweden. In total 134 neonates with extremely low birth weight (<1000g) and gestational age <28+0 weeks will be randomized to receive either dietary supplements of Lactobacillus reuteri or placebo. Study product will be identical to the active and placebo group besides the addition of Lactobacillus reuteri (1.25 x 100 million bacteria=0.2 ml oil drops per day) in the active group. The supplementation will commence within 1-3 days after birth and will be given daily until gestational week 36+0. The infants will be followed until gestational week 36+0 and data on feeding tolerance, nutrition, growth, infections, NEC, bronchopulmonary dysplasia, death, and potential confounders will be entered in an individual study protocol. Stool, breast milk, and blood samples will be collected for analyses of possible underlying mechanisms.

A 2-year follow up including examination by pediatrician, growth parameters, questionnaire and psychology testing (Bayley´s test) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight < 1000 g
* Gestational age: v23+0-V27 +6.
* Age < 72 hours at inclusion.
* Signed informed consent by parents.

Exclusion Criteria:

* Fatal or complex congenital malformation at inclusion time.
* Chromosomal defect at inclusion time.
* No realistic hope of survival at inclusion time.
* Gastrointestinal malformation at inclusion time.
* Participation in another study which aims to influence nutrition, growth, feeding tolerance or necrotizing enterocolitis.

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 134 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Abrahamsson, MD, PhD, Principal Investigator — Linköping University Hospital; County Council of Östergötland
Locations (2):
- Sweden (2):
  - Vrinnevi Hospital in Norrköping, Norrköping
  - Karolinska, Stockholm

REFERENCES:
- [Derived] Spreckels JE, Wejryd E, Marchini G, Jonsson B, de Vries DH, Jenmalm MC, Landberg E, Sverremark-Ekstrom E, Marti M, Abrahamsson T. Lactobacillus reuteri Colonisation of Extremely Preterm Infants in a Randomised Placebo-Controlled Trial. Microorganisms. 2021 Apr 24;9(5):915. doi: 10.3390/microorganisms9050915. PMID 33923278
- [Derived] Marti M, Spreckels JE, Ranasinghe PD, Wejryd E, Marchini G, Sverremark-Ekstrom E, Jenmalm MC, Abrahamsson T. Effects of Lactobacillus reuteri supplementation on the gut microbiota in extremely preterm infants in a randomized placebo-controlled trial. Cell Rep Med. 2021 Feb 22;2(3):100206. doi: 10.1016/j.xcrm.2021.100206. eCollection 2021 Mar 16. PMID 33763652

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Extremely preterm infants with a birth weight <1000 g were recruited within 72 hours after birth in two level 3 NICUs .
Pre-assignment Details: Inclusion should be completed to allow first dose of study product to be administered within 72 hours from birth.
Period: Overall Study
Arm/Group | Lactobacillus Reuteri | Placebo
Started | 68 | 66
Completed | 68 | 66
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Probiotic: Lactobacillus reuteri
- Total: Total of all reporting groups
Arm/Group | Probiotic | Placebo | Total
Number analyzed (Participants) | 68 | 66 | 134
Age, Continuous [Mean (Standard Deviation); unit: age in postmenstrual weeks at birth] — Postmenstrual weeks
  age in postmenstrual weeks at birth | 25.5 (1.2) | 25.5 (1.3) | 25.5 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 24 | 60
  Male | 32 | 42 | 74
Birth weight [Mean (Standard Deviation); unit: gram] | 731 (129) | 740 (148) | 735 (138)

OUTCOME MEASURES:

1. Primary Outcome: Time to Establish Full Enteral Feeds
Description: The age of the infants in days when the infant receive 150 ml/kg/day via enteral feeding for the first time.
Time Frame: Birth to gestational week 36+0
Population: Six infants - Four allocated to receive L. reuteri and two allocated to the placebo group died before reaching full enteral feeding and were not included in the analyses.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Lactobacillus Reuteri | Placebo
Number analyzed (Participants) | 64 | 64
days | 15 [11 to 23] | 15 [10 to 20]

2. Secondary Outcome: Days With Halted Feeding Due to Food Intolerance
Description: Episode with food intolerance. Retention volume> food volume given the last 2 hours (retention checked routinely every 4 hours) and/or clinical signs consistent with necrotizing enterocolitis (reduced general condition and inflated abdomen). The number of such events will also be indicated.
Time Frame: Birth to gestational week 36
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Lactobacillus Reuteri | Placebo
Number analyzed (Participants) | 68 | 66
days | 5.5 [3 to 9.5] | 6 [4 to 10]

3. Secondary Outcome: Number of Stools
Time Frame: Recorded over the first four weeks
Population: Only infants with complete records of stools during the first four weeks are included
Measure: Mean (95% Confidence Interval); unit: number of stools
Arm/Group | Lactobacillus Reuteri | Placebo
Number analyzed (Participants) | 47 | 44
number of stools | 69.6 [64.1 to 75.1] | 69.9 [63.8 to 75.9]

4. Secondary Outcome: Time Until Birth Weight is Regained. Specifies the Number of Full Days the Child Has Lived.
Description: Specifies the number of full days the child has lived.
Time Frame: Birth to gw 36+0
Reporting Status: Not Posted

5. Secondary Outcome: Weight Gain (SD)
Description: In this analysis, the difference in standard deviation score (delta z-scores) for weight, height and head circumference at birth and 14 and 28 days and gestational week 36+0 will be calculated. At gestational week 36+0 also absolute values will be analyzed. A positive delta z-score indicates faster growth than the growth chart would predict.
Time Frame: At 14th day of life
Measure: Mean (Standard Deviation); unit: change in standard deviations
Arm/Group | Lactobacillus Reuteri | Placebo
Number analyzed (Participants) | 64 | 62
change in standard deviations | -0.88 (0.81) | -0.88 (0.81)

6. Secondary Outcome: Mortality
Time Frame: Birth to gw 36+0
Measure: Number; unit: participants
Arm/Group | Lactobacillus Reuteri | Placebo
Number analyzed (Participants) | 68 | 66
participants | 5 | 5

7. Secondary Outcome: Necrotizing Enterocolitis
Description: Bell´s criteria II-III
Time Frame: Birth to gw 36+0
Measure: Number; unit: participants
Arm/Group | Lactobacillus Reuteri | Placebo
Number analyzed (Participants) | 68 | 66
participants | 7 | 8

8. Secondary Outcome: Sepsis
Description: Blood culture positive sepsis
Time Frame: Birth to gw 36+0
Measure: Number; unit: participants
Arm/Group | Lactobacillus Reuteri | Placebo
Number analyzed (Participants) | 68 | 66
participants | 25 | 23

9. Secondary Outcome: Bronchopulmonary Dysplasia
Description: Need of oxygen or CPAP/ventilator at gw 36+0
Time Frame: Gw 36+0
Population: Only patients surviving to gestational week 36+0 could be assessed for the diagnosis.
Measure: Number; unit: participants
Arm/Group | Lactobacillus Reuteri | Placebo
Number analyzed (Participants) | 63 | 61
participants | 40 | 39

10. Secondary Outcome: Weight Gain (SD)
Description: as for outcome 5
Time Frame: At 28th day of life
Measure: Mean (Standard Deviation); unit: change in standard deviations
Arm/Group | Lactobacillus Reuteri | Placebo
Number analyzed (Participants) | 64 | 63
change in standard deviations | -1.14 (1.07) | -1.25 (0.95)

11. Secondary Outcome: Weight Gain (SD)
Description: as for outcome 5
Time Frame: At gestational week 36+0
Measure: Mean (Standard Deviation); unit: change in standard deviations
Arm/Group | Lactobacillus Reuteri | Placebo
Number analyzed (Participants) | 63 | 61
change in standard deviations | -0.40 (1.30) | -0.24 (1.10)

12. Secondary Outcome: Length Gain (SD)
Description: as for outcome 5
Time Frame: At 14th day of life
Measure: Mean (Standard Deviation); unit: change in standard deviations
Arm/Group | Lactobacillus Reuteri | Placebo
Number analyzed (Participants) | 62 | 63
change in standard deviations | -1.02 (1.00) | -1.20 (1.01)

13. Secondary Outcome: Length Gain (SD)
Description: as for outcome 5
Time Frame: At 28th day of life
Measure: Mean (Standard Deviation); unit: change in standard deviations
Arm/Group | Lactobacillus Reuteri | Placebo
Number analyzed (Participants) | 62 | 62
change in standard deviations | -1.67 (1.47) | -1.96 (1.28)

14. Secondary Outcome: Length Gain (SD)
Description: as for outcome 5
Time Frame: At gestational week 36+0
Measure: Mean (Standard Deviation); unit: change in standard deviations
Arm/Group | Lactobacillus Reuteri | Placebo
Number analyzed (Participants) | 63 | 61
change in standard deviations | -1.44 (1.65) | -1.34 (1.52)

15. Secondary Outcome: Head Circumference Growth (SD)
Description: as for outcome 5
Time Frame: At 14th day of life
Measure: Mean (Standard Deviation); unit: change in standard deviations
Arm/Group | Lactobacillus Reuteri | Placebo
Number analyzed (Participants) | 61 | 62
change in standard deviations | -0.92 (0.56) | -1.11 (0.82)

16. Secondary Outcome: Head Circumference Growth (SD)
Description: as for outcome 5
Time Frame: At 28th day of life
Measure: Mean (Standard Deviation); unit: change in standard deviations
Arm/Group | Lactobacillus Reuteri | Placebo
Number analyzed (Participants) | 64 | 63
change in standard deviations | -1.21 (0.85) | -1.73 (0.91)
Statistical Analysis 1: Comparison: Lactobacillus Reuteri vs Placebo; Test type: Other — Student's t-test; p = 0.001, t-test, 2 sided

17. Secondary Outcome: Head Circumference Growth (SD)
Description: as for outcome 5
Time Frame: At gestational week 36+0
Measure: Mean (Standard Deviation); unit: change in standard deviations
Arm/Group | Lactobacillus Reuteri | Placebo
Number analyzed (Participants) | 63 | 61
change in standard deviations | -0.57 (1.29) | -0.79 (1.24)

18. Secondary Outcome: Neurological Development
Description: Bayleys´s test by psychologist
Time Frame: At 2 years corrected age
Reporting Status: Not Posted, anticipated posting 2024-08

19. Secondary Outcome: Neurological Development Impairment
Description: A composite of several outcomes: impaired cognition at the Bayleys´test, cerebral palsy, blindness and deafness, divided into normal, mild, moderate and severe. Mild -1SD to -2SD, Moderate <-2D to 3 SD and Severe <3SD
Time Frame: At 2 years corrected age
Reporting Status: Not Posted, anticipated posting 2024-08

ADVERSE EVENTS:
Time Frame: From birth until 36+0 weeks corrected postmenstrual age
Arm/Group | Lactobacillus Reuteri | Placebo
All-Cause Mortality (participants affected / at risk) | 5/68 | 5/66
Serious Adverse Events (participants affected / at risk) | 55/68 | 52/66
Other Adverse Events (participants affected / at risk) | 0/68 | 0/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lactobacillus Reuteri (N=68) | Placebo (N=66)
Infection by the probiotic bacterium (Infections and infestations) | 0 (0) | 0 (0) — Positive culture with Lactobacillus reuteri from a normally sterile location (typically blood, cerebrospinal fluid).
Severe morbidity or death (General disorders) | 55 | 52 — This compound measure reports if any of the following occurred: Necrotizing enterocolitis stage 2 - 3 Culture proven sepsis Bronchopulmonary dysplasia ROP, grade 3-5 IVH, grade 3-4 Periventricular leukomalacia Death

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No